CLINICAL TRIAL: NCT01260571
Title: Clinical Study to Evaluate the Efficacy of Topical Medications Containing Benzoyl Peroxide and Sulfur in the Regression in the Short Time (24 Hours) of Moderate Acne Vulgaris Grade II (Pimples)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zurita Laboratorio Farmaceutico Ltda. (Industry)
Responsible Party: Sergio Schalka, Medicin Skin Institute
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EAA 554-10/v6
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-09

CONDITIONS: Treatment of Acne Vulgaris Grade II in a Short Period of Time.
Keywords: blackheads and pimples; Acne vulgaris grade II
MeSH Terms: interventions — Benzoyl Peroxide; Sulfur

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Benzoyl Peroxide and Sulfur (Experimental): Topical Medications containing benzoyl peroxide and sulfur
  Interventions: Drug: Benzoyl peroxide and sulfur

INTERVENTIONS:
Drug: Benzoyl peroxide and sulfur — topical cream, 5% benzoyl peroxide and 2% sulfur Frequency once to day Duration 24 hours

SUMMARY:
Sixty two subjects will take part in this study. The study is unic arm. The subjects used the product once and will be evaluated in the regression of pimples in the times 0,4,6,8 and 24 hours after application.

A follow-up visit will be made 24 hours after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes aged to 12 years to 35 years
* Oily skin prone to acne
* Presence of at least three inflammatory lesions, diagnosed as grade II acne vulgaris.
* Sign the informed Consent Form
* Comply the requirements and attend to study visits

Exclusion Criteria:

* Pregnancy (need for urinary pregnancy test for women of childbearing age)
* Lactation
* Presence of acne conglobata and nodulocystic
* Pathologies associated hormonal (thyroid diseases, ovaries micropolycystic)
* Drug use systemic corticosteroids, anticonvulsants and / or new drugs for up to one month before to selection.
* History of atopy or allergic cutaneous
* History of hypersensitivity to benzoyl peroxide and sulfur
* Beginning or ending the use of contraceptives (for females)
* Intense sun exposure until one month before the evaluation

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Clinical study to evaluate the efficacy of topical medications containing benzoyl peroxide and sulfur in the regression in the short time (24 hours) of moderate acne vulgaris grade II (pimples). | 24 hours
  Clinical evolution of the target lesions for each experimental time regarding the parameters of reddening, size and general appearance of the lesion.

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele, Osasco, São Paulo, Brazil